CLINICAL TRIAL: NCT00515164
Title: Phase 2 Study of the 20 mL Biologic Lung Volume Reduction System (BLVR) in Patients With Advanced Upper Lobe Predominant Emphysema
Brief Title: US Biologic Lung Volume Reduction (BLVR) Phase 2 Emphysema Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-C07-001
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Pulmonary Emphysema; Chronic Obstructive Pulmonary Disease
Keywords: lung volume reduction; emphysema; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Emphysema; Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Hydrogels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Treatment will be administered in 2 treatment sessions.
  Interventions: Drug: Biologic Lung Volume Reduction (BLVR) - 20 mL Hydrogel
- Group 2 (Experimental): Treatment will be administered in a single treatment session.
  Interventions: Drug: Biologic Lung Volume Reduction (BLVR) - 20 mL Hydrogel

INTERVENTIONS:
Drug: Biologic Lung Volume Reduction (BLVR) - 20 mL Hydrogel — 20 mL Hydrogel

SUMMARY:
The purpose of this study it to evaluate the efficacy and safety of the 20 mL BLVR System in patients with advanced upper lobe predominant emphysema.

DETAILED DESCRIPTION:
Background:

Patients with emphysema currently have limited treatment choices. Many patients are treated with steroids and inhaled medications, which often provide little or no benefit. In recent years, lung volume reduction surgery has become an accepted therapy for advanced emphysema. Lung volume reduction surgery involves the removal of diseased portions of the lung in order to enable the remaining, healthier portions of the lung to function better. This procedure, although effective for many patients, is complicated and is accompanied by substantial morbidity and mortality risk.

Aeris Therapeutics has developed the Biologic Lung Volume Reduction (BLVR) System which is intended to achieve lung volume reduction without surgery and its attendant risks. Patients are treated using a bronchoscope to direct treatment to the most damaged areas of the lung. The treatment delivers a precisely proportioned proprietary mixture of drugs and biologics which, when combined at the treatment site, form a biodegradable hydrogel. The hydrogel acts to reduce lung volume by permanently collapsing and sealing the diseased areas of the lung. This provides room within the chest to allow the remaining healthier portions of the lung to function better.

Aeris' BLVR development program has been granted Fast Track designation by the U.S. FDA, and is the subject of ongoing clinical trials designed to investigate the safety and efficacy of the BLVR System as a treatment for patients with advanced heterogeneous emphysema. Fast Track designation is reserved for drug and biologic development programs that are intended to treat serious or life-threatening conditions and that demonstrate the potential to address unmet medical needs.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of advanced upper lobe emphysema
* age >/= 40 years
* clinically significant dyspnea
* failure of standard medical therapy to relieve symptoms (inhaled beta agonist & inhaled anticholinergic)
* pulmonary function tests within protocol-specified ranges (post bronchodilator FEV1 < 45% predicted & experiencing < 30% or 300 mL improvement using bronchodilator; total lung capacity > 110% predicted; residual volume > 150% predicted)
* 6 Minute Walk Distance >/= 150 m

Exclusion Criteria:

* alpha-1 protease inhibitor deficiency
* homogeneous emphysema
* tobacco use within 4 months of initial visit
* body mass index < 15 kg/m2 or> 35 kg/m2
* clinically significant asthma, chronic bronchitis or bronchiectasis
* allergy or sensitivity to procedural components
* pregnant, lactating or unwilling to use birth control if required
* prior lung volume reduction surgery, lobectomy, pneumonectomy, lung transplant, endotracheal valve placement, airway stent placement or pleurodesis
* comorbid condition that could adversely influence outcomes
* inability to tolerate bronchoscopy under conscious sedation (or anesthesia)
* history of renal infarction or renal failure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Reduction in gas trapping | 12 weeks post treatment
SAEs - Safety of treatment and the procedure | 2 years post treatment

SECONDARY OUTCOMES:
Improvement in exercise capacity | 12 weeks post treatment
Improvement in vital capacity | 12 weeks post treatment
Improvement in expiratory flow | 12 weeks post treatment
Improvement in inspiratory flow | 12 weeks post treatment
Improvement in dyspnea symptoms (breathlessness) | 12 weeks post treatment
Improvement in respiratory quality of life | 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey McLennan, MD, Principal Investigator — University of Iowa Hospitals & Clinics, Iowa City, IA; Charlie Strange, MD, Principal Investigator — Medical University of South Carolina; Mark Gotfried, MD, Principal Investigator — Pulmonary Associates, Phoenix, AZ; Mark Krasna, MD, Principal Investigator — St Joseph's Medical Center, Towson, MD; Sanjiv Tewari, MD, Principal Investigator — Akron Medical Center, Akron, OH; Gerard Criner, MD, Principal Investigator — Temple University Lung Center, Philadelphia, PA; William Leeds, DO, Principal Investigator — Veritas Clinical Specialties, Topeka, KS; Thomas Gildea, MD, Principal Investigator — Pulmonary, Allergy & Critical Care Medicine, Cleveland Clinic, Cleveland, OH
Locations (8):
- United States (8):
  - Pulmonary Associates, Phoenix, Arizona
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Veritas Clinical Specialties, Ltd, Topeka, Kansas
  - St Joseph's Medical Center, Towson, Maryland
  - Akron Medical Center, Akron, Ohio
  - Pulmonary, Allergy & Critical Care Medicine, Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple University Lung Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Background] Ingenito EP, Berger RL, Henderson AC, Reilly JJ, Tsai L, Hoffman A. Bronchoscopic lung volume reduction using tissue engineering principles. Am J Respir Crit Care Med. 2003 Mar 1;167(5):771-8. doi: 10.1164/rccm.200208-842OC. Epub 2002 Oct 11. PMID 12406835
- [Background] Reilly J, Washko G, Pinto-Plata V, Velez E, Kenney L, Berger R, Celli B. Biological lung volume reduction: a new bronchoscopic therapy for advanced emphysema. Chest. 2007 Apr;131(4):1108-13. doi: 10.1378/chest.06-1754. PMID 17426216
- [Derived] Criner GJ, Pinto-Plata V, Strange C, Dransfield M, Gotfried M, Leeds W, McLennan G, Refaely Y, Tewari S, Krasna M, Celli B. Biologic lung volume reduction in advanced upper lobe emphysema: phase 2 results. Am J Respir Crit Care Med. 2009 May 1;179(9):791-8. doi: 10.1164/rccm.200810-1639OC. Epub 2009 Jan 29. PMID 19179484